CLINICAL TRIAL: NCT05615246
Title: An Open Label, Multi-Center, Retrospective and Prospective Evaluation of Exactech Humeral Reconstruction Prosthesis of Shoulder Arthroplasty
Brief Title: Exactech Humeral Reconstruction Prosthesis of Shoulder Arthroplasty PMCF (HRP)
Acronym: HRP
Status: Terminated | Type: Observational
Why Stopped: Site closeout
Sponsor: Exactech (Industry)
Responsible Party: Sponsor
Other Study IDs: CR18-001
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis Shoulder; Rheumatoid Arthritis; Oncology
MeSH Terms: conditions — Arthritis, Rheumatoid; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to collect and evaluate long-term clinical outcomes data in order to better understand the safety and performance of the Equinoxe Humeral Reconstruction Prosthesis in shoulder arthroplasty over time. This study will follow subjects for a period of up to 10 years post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient is indicated for shoulder arthroplasty (or has previously undergone shoulder arthroplasty)
* Patient is at least 21 years of age
* Patient is expected to survive at least 2 years beyond surgery
* Patient is willing to participate by complying with pre- and postoperative visit requirements
* Patient is willing and able to read and sign a study informed consent form

Exclusion Criteria:

* Osteomyelitis of the proximal humerus or scapula; if a systemic infection or a secondary remote infection is suspected or confirmed, implentation should be delayed until infection is resolved
* Inadequate or malformed bone that precludes adequate support or fixation of the prosthesis
* Neuromuscular disorders that do not allow control of the joint
* SIgnigicant injury to the brachial plexus
* Non-functional deltoid muscles
* Patient's age, weight, or activity level would cause the surgeon to expect early failure of the system
* The patient is unwilling or unable to comply with the post-operative care instructions
* Alcohol, drug, or other subtance abuse
* Any disease state that could adversely affect the function or longevity of the implant
* Patient is pregnant
* Patient is a prisoner
* Patient has a physical or mental condition that would invalidate the results

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients who meet eligibility criteria
  * Patients who consent to participate to return for follow-up visits out to 10 years or longer
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
SST-12 | Through study completion, an average of 1 per year
  Shoulder Simple Test (SST) - 12 questions with yes/no responses that measure shoulder pain and function from a patient's perspective - 12 yes corresponds to 100%
SPADI | Through study completion, an average of 1 per year
  Shoulder Pain and Disability Index (SPADI) -13 questions assessing about pain scale (5 questions) and disability scale (8 questions) where 0 indicates no pain/no difficulty and 10 indicates worst pain imaginable/so difficult it requires help while performin these activities
Constant | Through study completion, an average of 1 per year
  Constant Shoulder Score - 100 points scale about pain, Activities of daily living, Strength test, and Range of Motions questions about shoulder where 100 % corresponds to the highest pain
ASES | Through study completion, an average of 1 per year
  American Shoulder and Elbow Surgeons Score (ASES) - 100 points scale about shoulder pain and performance evaluation in activities of daily living where 100 indicates the best shoulder condition
UCLA | Through study completion, an average of 1 per year
  University of California Los Angeles Shoulder Score (UCLA) - 5 Items score which combines both physician (3 items) and patient assessment (2 items) whith a total range from 0-35 where 0 indicates worse shoulder function and 35 better shoulder function outcomes
TESS | Through study completion, an average of 1 per year
  Toronto Extremity Salvage Score (TESS) - Patient functional assessment following for surgery for musculoskeletal tumors (Humeral Reconstruction Stem only) - 100-point score where higher score indicates a better outcome
MSTS | Through study completion, an average of 1 per year
  Musculoskeletal Tumor Society (MSTS) - 30 points [6 times (range 0-5)], simple measure of the upper extremity function (Humeral Reconstruction Stem only) - The maximum corresponds to the best score

CONTACTS AND LOCATIONS:
Locations (1):
- Western Orthopaedics Research and Education Foundation, Denver, Colorado, United States